CLINICAL TRIAL: NCT01415986
Title: Interstitial Photodynamic Therapy (PDT) With Temoporfin for Advanced Head and Neck Cancers - PHASE II PILOT STUDY
Brief Title: Interstitial Photodynamic Therapy (PDT) With Temoporfin for Advanced Head and Neck Cancers
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The patient was "lost to follow-up" and the PI left the institution.
Sponsor: University of Arkansas (Other)
Collaborators: Erasmus Medical Center (Other); The Netherlands Cancer Institute (Other); Biolitec Pharma Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UAMS IRB 114294
Record Dates: First submitted 2011-08-10; First posted 2011-08-12 (Estimated); Results first posted 2012-12-03 (Estimated); Last update posted 2012-12-03 (Estimated); Status verified 2012-11

CONDITIONS: Squamous Cell Carcinoma of the Head and Neck
Keywords: Advanced head and neck cancer; Squamous cell carcinoma; SCC; HNSCC
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck; Head and Neck Neoplasms; Carcinoma, Squamous Cell | interventions — temoporfin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Subjects receiving Temoporfin (Experimental)
  Interventions: Drug: Temoporfin; Device: Medical diode laser emitting light at a wavelength of 652 nm. (Ceralas PDT 652, CeramOptec GmbH)

INTERVENTIONS:
Drug: Temoporfin — A single dose of 0.15 mg of Temoporfin per kilogram of body weight will be administered by slow intravenous injection into a deep vein (such as the antecubital vein) in not less than 6 minutes.
  Other Names: Foscan
Device: Medical diode laser emitting light at a wavelength of 652 nm. (Ceralas PDT 652, CeramOptec GmbH) — Light dose of 20 J/cm, at a rate of 100 mW/cm, will be delivered to the target tumor and margins, within 200 seconds.
  Other Names: Ceralas PDT 652, CeramOptec GmbH

SUMMARY:
Presently, there is no effective treatment for patients with advanced head and neck cancer (AHNC) that failed to respond to the standard therapy (radiation, chemotherapy and surgery) in the US. These patients are deemed incurable AHNC. In the European Union (EU), interstitial photodynamic therapy (I-PDT) with Temoporfin is approved for the treatment of patients with incurable AHNC. Well designed EU studies have shown that I-PDT with Temoporfin can provide worthwhile palliation by reducing tumor size, bleeding and pain in 53% - 60% of patients with incurable AHNC. This is a significantly higher rate in comparison to the reported response rate of palliative chemotherapy (6-30%). However, the EU studies did not correlate quantitative tumor response with clinical outcome. In addition, quality of life (QoL) improvements associated with I-PDT of AHNC using Temoporfin were also not evaluated.

The objective of this study is to quantify the tumor response and patient's QoL to I-PDT with Temoporfin. Successfully meeting this objective will give us the tools the investigators need to design larger studies to significantly improve the management and QoL of patients with AHNC.

DETAILED DESCRIPTION:
This is a non-randomize, open label, Pilot phase II study with 5 consenting subjects. The specific aims of this study are:

Aim 1: Quantitate local tumor response in patients with incurable AHNC treated with I-PDT with Temoporfin.

Aim 2: Evaluate the changes in QoL in patients with incurable AHNC treated with I-PDT with Temoporfin.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age and older, male or female, of all races and ethnicities.
* Prior histologically confirmed advanced squamous cell carcinoma of the head and neck that failed standard therapy (radiation, chemotherapy, surgery).
* Must have a Karnofsky performance status higher than 70%.
* Measurable disease by PET-CT, defined as maximum SUV ≥4 in FDG for the tumor.
* Must have a discrete tumor that is accessible for unrestricted illumination of interstitial photodynamic therapy (I-PDT).
* Deemed unsuitable, by multidisciplinary tumor board, for curative treatment options such as radiotherapy, surgery, chemotherapy or a combination of these modalities. This will include patients who have exceeded the maximum radiation dose and are not candidates for re-irradiation.
* Deemed likely to survive for at least 6 months.
* Able and willing to provide written informed consent to participate in the study.
* If a female of childbearing potential, the subject is willing to take a pregnancy test and practice strict birth control (estrogen-containing oral contraceptives or an intrauterine device) throughout the study and for 3 months after Temoporfin administration. Women who have had a hysterectomy are exempt from these requirements.
* Must have blood glucose level below 250 (and preferably below 200) before FDG injection, required for PET-CT.
* Willing to remain in a light-avoidance environment for a time period of at least 15 days.
* Laboratory criteria:

  * Hematocrit >= 33%, hemoglobin >= 11 g/dl
  * Platelet count >70.000 per microliter
  * BUN: 7 to 20 mg/dL
  * CO2 (carbon dioxide): 20 to 29 mmol/L
  * Creatinine: 0.8 to 1.4 mg/dL
  * Glucose: 64 to 128 mg/dL
  * Serum chloride: 101 to 111 mmol/L
  * Serum potassium: 3.7 to 5.2 mEq/L
  * Serum sodium: 136 to 144 mEq/L
  * Liver function test: albumin, bilirrubin (direct/conjugated), ALT (alanine transaminase), AST (aspartate transaminade), GGT (gamma glutamyl transferase), ALP (alkaline phosphatase) within normal limits
  * White blood count > 3,000 per microliter or ANC > 1500 per microliter
  * Serum calcium within normal limits.

Exclusion Criteria:

* A tumor that is too close to a major blood vessel (such as the carotid artery).
* A tumor invading the skull base.
* The tumor is not clearly shown on the CT image.
* The location and extension of the tumor precludes an effective I-PDT.
* Pregnant or has uncontrolled hyperglycemia.
* Has porphyria or other diseases exacerbated by light.
* With hypersensitivity to Temoporfin or to any of its excipients.
* Has known allergies/hypersensitivity to porphyrins.
* Has known sensitivity to the CT contrast agent. (Omnipaque)
* Has poor renal function as demonstrated by serum creatinine and EGFR <40, which would preclude the using of the CT contrast agent.
* Patient with a planned surgical procedure within the next 30 days.
* Has a coexisting ophthalmic disease likely to require slit-lamp examination within the next 30 days.
* Patient with existing therapy with a photosensitizing agent (Temoporfin, protoporphyrin or derivatives of porphyrin).
* Has received prior photodynamic therapy to the proposed treatment site within the prior 3 months.
* Has distant metastasis (with the exception of single stable distant metastasis that does not decrease life expectancy to less than 6 months).
* Has a childbearing potential and will not use adequate contraceptive protection.
* A female that is breastfeeding.
* Patient of childbearing potential who has a positive (+) urine pregnancy test.
* Received treatment with an experimental drug or entered another clinical trial within the prior 30 days.
* Received radiotherapy to the head and neck region within the prior 3 months.
* Any disease, which is caused or exacerbated by light, including systemic lupus erythematosus, psoriasis, porphyria, actinic reticuloid or xeroderma pigmentosum.
* Has been treated within the prior 30 days with a light-activated therapy or other medication that may render the subject photosensitive (e.g., psoralen ultraviolet A-range [PUVA], Accutane, 5-Fluorouracil, tetracycline's ).
* Not willing or able to complete the visit requirements of this protocol or adhere to the instructions regarding light exposure.
* Any other condition that the PI staff feels will be an endangerment to the subject.

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2010-11; Primary Completion 2011-08 (Actual); Study Completion 2012-03 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Arkansas for Medical Sciences, Little Rock, Arkansas, United States

REFERENCES:
- [Background] Lou PJ, Jager HR, Jones L, Theodossy T, Bown SG, Hopper C. Interstitial photodynamic therapy as salvage treatment for recurrent head and neck cancer. Br J Cancer. 2004 Aug 2;91(3):441-6. doi: 10.1038/sj.bjc.6601993. PMID 15238981

RESULTS

PARTICIPANT FLOW:
Groups:
- Group 1: Interstitial Photodynamic Therapy (I-PDT). This subject was adminatred with 0.15 mg/kg Foscan on day 1. He was trtaed with I-PDT using 652-nm light at 20 J/cm, 4 days after the drug adminstration. He stayed in a outpatient facility for 3 more days and discharged home.
Period: Overall Study
Arm/Group | Group 1
Started | 1
Completed | 0 (Study terminated)
Not Completed | 1
Not completed — Lost to Follow-up | 1

BASELINE CHARACTERISTICS:
Groups:
- Group 1: Interstitial Photodynamic Therapy (I-PDT)
Arm/Group | Group 1
Number analyzed (Participants) | 1
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 0
  >=65 years | 1
Age Continuous [Mean (Standard Deviation); unit: years] | 65 (0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 1
Region of Enrollment [Number; unit: participants]
  United States | 1

OUTCOME MEASURES:

1. Primary Outcome: Local Tumor Response to Interstitial Photodynamic Therapy (I-PDT) With Temoporfin
Description: Longitudinal changes in tumor size (cm) and standardized uptake value (SUV) measured with Positron Emission Tomography - Computed Tomography (PET- CT).
Time Frame: Within 1 month of enrollment or as scheduled at screening and at 3 and 5 months after treatment
Population: No data was collected because the participant was lost to follow up.
Groups:
- Group 1: Interstitial Photodynamic Therapy (PDT)
Arm/Group | Group 1
Number analyzed (Participants) | 0

2. Secondary Outcome: Changes in the Quality of Life (QoL)
Description: The change in the overall score of the University of Washington quality of life questionnaire (UW-QOL). Each of the domain-specific items is scored from 0 (worst quality of life (QOL) to 100 (Best QOL). The composite score is created by averaging the scores.
Time Frame: Within 1 month of enrollment or as scheduled at screening and at 3 and 5 months after treatment.
Population: No data was collected because the participant was lost to follow up.
Arm/Group | Group 1
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Arm/Group | Group 1
Serious Adverse Events (participants affected / at risk) | 1/1
Other Adverse Events (participants affected / at risk) | 0/1
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1 (N=1)
Death (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) — The subject death was due to the natural course of the disease. Not related to the study.

LIMITATIONS AND CAVEATS:
Early termination leading to small numbers of subjects analyzed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No